CLINICAL TRIAL: NCT06419868
Title: Acceptability and Feasibility of a Universal Preventive Intervention for Depression and Anxiety in University Students
Brief Title: Acceptability and Feasibility of a Universal Preventive Intervention
Acronym: FDI2024
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Tenured Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FDI UAN23102
Record Dates: First submitted 2024-04-30; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Depression/Anxiety
Keywords: Depression; Anxiety; Undergraduates; Universal prevention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is an experimental study, with a randomized controlled trial design, with a control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This is a self-applied online intervention with six modules. It should be implemented over a period of 4 to 8 weeks. Participants will be guided through the program in a structured manner. They will start by accessing the CANVAS online platform, where they will find the content of the sessions in video, audio, and text formats. They will then be directed to practice exercises at home, with audiovisual material to guide them. It's crucial that participants complete the six sessions sequentially, as each session is designed to build upon the previous one, ensuring a comprehensive learning experience and effective learning.
  Interventions: Behavioral: "Universal preventive intervention for depression and anxiety for university students"
- Control group (No Intervention): Control group participants will be asked to respond to the baseline, after intervention, and four months after intervention. Once the study period is completed, and if the results show positive changes in the intervention group, they will be offered and asked to access the intervention.

INTERVENTIONS:
Behavioral: "Universal preventive intervention for depression and anxiety for university students" — This is a self-applied online intervention with six modules. It should be implemented over a period of 4 to 8 weeks. It includes emotion regulation, mindfulness exercises, coping strategies, problem-solving strategies, psychoeducation of anxiety and depression, and the development of healthy behaviors, explained through the following theoretical components: mindfulness and cognitive behavioral therapy.
  Participants will be guided through the program in a structured manner. They will start by accessing the CANVAS online platform, where they will find the content of the sessions in video, audio, and text formats. They will then be directed to practice exercises at home, with audiovisual material to guide them. It's crucial that participants complete the six sessions sequentially, as each session is designed to build upon the previous one, ensuring a comprehensive learning experience and effective learning.
  Other Names: Cuidate
  Arms: Intervention group

SUMMARY:
Mental health in the university population has become a common and serious problem within university institutions worldwide in recent years. Various meta-analyses and systematic reviews have shown worrying figures in the last five years. In the USA, it has been described in medical students that between 6.0% and 66.5% have depression, between 7.7% and 65.5% anxiety disorders, and between 12.2% and 96.7% present stress. In China, on the other hand, a study reported in 2016 that the prevalence of depression was 23.8%. In Latin America, a Brazilian article conducted on medical students shows a prevalence of depression at 30.6%, anxiety disorders at 32.9%, and stress at 49.9%.

In Chile, there are very few studies that address the prevalence of mental health disorders and associated risk factors in the university population. The article published in 2014 by Baader et al. is one of the first records was carried out on a population of 800 students in 2008 at the Austral University of Chile, reporting a prevalence of 27% of depression and 5.3% of students who present a moderate to severe risk of suicide. During April and May 2019, the results of the "First National University Mental Health Survey" project were presented, a project led by the Catholic University of Temuco and sponsored by the National Research and Development Agency (ANID), carried out to 600 students from the Catholic University of Temuco, the University of Concepción and the University of Tarapacá. This project showed that 46% of the students presented depressive symptoms, 46% anxiety symptoms, and 53.5% stress symptoms. Furthermore, 29.7% presented the three symptoms simultaneously, and 5.1% of the students had suicidal thoughts at the time of the study.

In a review of published studies on mental health in higher education students in Chile, a wide variability in the prevalence of psychological symptoms among students was identified. The findings showed a range of prevalence of psychological distress between 22.9% and 40.7%, of depressive symptoms between 16.5% and 38.8%, of anxious symptoms between 16.5% and 23.7%, of cannabis consumption in the last 12 months between 19.7% and 29.7%, and alcohol consumption in the previous year between 84.0% and 92.6%.

The data obtained from the Mental Health Surveys of the University of the Andes, applied in the years 2020 and 2022 to undergraduate students, indicate variations in the prevalence of different symptoms and psychological risks. Specifically, the prevalence of depressive symptoms decreased from 37.1% to 27.84%, and that of anxious symptoms decreased slightly from 37.9% to 36.13%. A notable decrease was observed in stress, going from 54.6% to 12.9%. On the other hand, the prevalence of suicide risk experienced a less pronounced decrease, from 20% to 18.4%, remaining at a considerably high rate.

Taking into account the above, mental health problems in the university population continue to be a public health problem that must be addressed preventively through the implementation of evidence-based programs.

Objective: This study aims to determine the acceptability and feasibility of an online universal mental health prevention program for university students. It is also expected to reduce depressive and anxious symptoms and improve quality of life.

Outcomes:

Primary response measures: Acceptability Assessment, Feasibility Assessment. Secondary response measures are depression, anxiety, and quality of life. The Outcomes section provides more details on anxiety and qu.

Expected results: The data collected will allow us to determine the acceptability and satisfaction of the participants with the intervention using a quantitative measure of its credibility and to explore its effects on the participants, considering the change in depressive and anxiety symptoms and quality of life before and after the intervention.

DETAILED DESCRIPTION:
STRATEGIES AND INTERVENTIONS ORIENTED ON THE PROMOTION AND PREVENTION OF MENTAL HEALTH PROBLEMS:

Recent research highlights the effectiveness of preventive interventions on the mental health of university students, whether through digital media, in-person actions, or a combination of both. The contents of these interventions have allowed us to establish the mechanisms and main mediators that explain the effectiveness of these interventions. For example, recent studies have demonstrated the positive effects of mindfulness on individual health, decreasing the intensity of distress, accelerating emotional recovery, and increasing the ability to engage in goal-oriented behavior. In mindfulness training, people learn to self-regulate their attention. In this sense, in 2021, a pilot study with a control group was carried out at the Universidad de los Andes (ClinicalTrials.gov Identifier: NCT05114824) in which an intervention based on Mindfulness with cognitive-behavioral elements of 8 sessions was evaluated in undergraduate students. It showed a significant reduction in depressive and anxiety symptoms and an increase in quality of life in those students who participated in the intervention compared to the control group. This intervention was based on a program developed by Dr. Elizabeth English and evaluated by Dr. Julieta Galante at the University of Cambridge with excellent results. Another study in England evaluated a mindfulness intervention, which achieved notable reductions in perceived stress (d = -1.25), anxiety (d = -1.09), and depression (d = -1.06) in comparison with a control group, with sustained benefits during 3 and 6 month follow-ups.

In Germany, a study evaluated an Internet-based intervention supported by a mobile application called "StudiCareStress." This intervention is based on cognitive-behavioral and third-wave techniques. It aligns with Lazarus' transactional model of stress by differentiating between problem-focused coping and coping focused on emotion regulation. Cognitive-behavioral problem-solving strategies are applied for problem-focused coping to reduce and eliminate modifiable stressors. Emotion regulation is how individuals monitor, evaluate, modify, and manage emotions to achieve relevant needs or goals. It has been shown to influence the reduction of various symptoms of emotional distress. The intervention comprised eight main modules. Completing 1 module took 30 to 90 minutes, and participants were recommended to complete at least one and a maximum of 2 modules per week. Therefore, the intervention was intended to be completed in approximately 5 to 7 weeks. This study revealed significant effects on stress relief (d = 0.69), anxiety (d = 0.76), depression (d = 0.63), and improvements in academic productivity (d = 0.33). ) and academic work performance (d = 0.34) after seven weeks.

Another study in Australia evaluated the "moodgym" program, a program that is delivered over the Internet and is entirely self-administered. This program incorporates cognitive behavioral strategies such as "attentional bias modification" and "information processing." About the modification of attention bias, they are strategies that reduce the tendency of individuals with emotional disorders to pay too much attention to negative information. These strategies enable people to reduce attention to this negative information but, at the same time, actively use positive or neutral information. On the other hand, "information processing" strategies try to reduce the biases that can occur in individuals with emotional disorders such as depression, on the one hand, disconnect from negative content, improve the processes of information interpretation, and reduce memory biases. Participants completed the intervention for six weeks in the study that evaluated this program. Participants were asked to spend 40 minutes weekly on "moodgym", complete the sessions in one sitting, and only log into "moodgym" when prompted. Participants who completed the intervention had continued improvement in depressive symptoms. Furthermore, significantly fewer people in the intervention condition had diagnostic criteria for major depression at follow-up than in the control group.

In a recent review, it was concluded that Internet-based interventions for the mental health of university students can have significant effects on depression, anxiety, and other mental health problems. When reviewing the components of the programs included in this review, it was also possible to conclude that the majority of these interventions, in addition to incorporating training in specific skills, either from cognitive behavioral theory or different aspects of emotional regulation, most of them also incorporate psychoeducational aspects and others related to the development of healthy behaviors such as the use of physical exercise and sleep hygiene.

Unfortunately, in Chile and Latin America, no studies have evaluated preventive interventions using technology in the university population. All the results presented come from developed countries, but they are guidelines when designing an intervention that could be effective in our context. It is also important to mention that whatever the intervention, it must, on the one hand, incorporate the components that have been demonstrated as mediators in the prevention of depression and anxiety. On the other hand, they should be culturally relevant to promote involvement and adherence to this type of intervention in the university population. Whether through an internet platform or mobile applications, technology-based interventions are very promising in facilitating students' access to this content. In particular, the Universidad de los Andes has a CANVAS platform that favors students' work in their regular academic activities. Based on the experience shown in other interventions, such as the "moodgym" intervention, it can be expected that if these platforms are culturally attractive to students, they can generate better adherence. Finally, technology allows us to get closer to the common language in which university students are immersed. At the same time, if these interventions are effective, they have a high potential for scaling up to promote better well-being at the population level. These underscore the effectiveness of technology-based interventions, not only in improving mental health symptoms but also in the accessibility and appeal of these programs to students who might not otherwise seek help.

Based on the above review, a successful universal mental health prevention program for university students should incorporate strategies that promote emotion regulation, a crucial component for well-being and social adaptation. Integrating mindfulness techniques and cognitive-behavioral therapy would make it easier for individuals to recognize and adequately manage their emotions. Likewise, the literature suggests the importance of developing skills for coping with academic stress through effectively assessing stressful situations and implementing strategies focused on problem-solving and emotional regulation skills. In addition, and according to the review, aspects of psychoeducation on stress, anxiety and depression, problem-solving, and development of healthy behaviors, such as physical activity and sleep care, should also be incorporated.

In this study, the principal investigator propose to develop and evaluate a brief online intervention that incorporates the mediators of effectiveness demonstrated in other interventions, such as training in mindfulness skills, emotional regulation, coping with academic stress, problem-solving, and interpersonal effectiveness, which will prevent symptoms of depression and anxiety on undergraduate students.

2. Objectives: This study aims to determine the acceptability and feasibility of an online universal mental health prevention program for university students. It is also expected to reduce depressive and anxious symptoms and improve quality of life.

2.1. Primary objectives

1. Develop an online intervention aimed at preventing depression and anxiety, strengthening emotional regulation skills, mindfulness techniques, healthy coping with stress, problem-solving, psychoeducational skills, and healthy behaviors.
2. Determine the participant's acceptability and satisfaction with the intervention using the Client Satisfaction Questionnaire (CSQ-8).
3. Determine the feasibility of recruiting study subjects, retaining participants, attending sessions, and collecting quantitative data during the program.

2.2. Secondary objectives

(1) Evaluate the effects of the intervention on the participants, their depressive and anxious symptoms, and their quality of life.

3. Design: This experimental study has a randomized controlled trial design and a control group.

4. Participants: The participants will be undergraduate students from the Universidad de los Andes with different majors.

5. Intervention: There are no proven interventions in university students that have evidence in Chile, but the literature review highlights interventions that have worked in countries such as England, Germany and Australia, which incorporate the following contents and mediators: emotion regulation, mindfulness techniques, coping skills, problem-solving, psychoeducation of anxiety and depression and development of healthy behaviors. In this project, the principal investigator will propose the design and creation of a self-applied online intervention that incorporates these components, and that should initially have six modules, which should be implemented in 4 to 8 weeks. Participants will receive access to the CANVAS platform, where they will find the sessions' content in video, audio, and text format. In addition, they will be asked to practice some techniques at home, with audiovisual material to guide them. Participants will be asked to complete the six sessions sequentially, completing each one before advancing to the next. Session attendance data will be collected and evaluated.

6. Outcomes: 6.1. Primary response measures 6.1.1. Acceptability Assessment Acceptability will be evaluated by determining how this intervention program is received by students and the extent to which this intervention relates to the needs of this target population. At the end of the program, the research team will develop an acceptability and satisfaction questionnaire for the intervention students. In addition, the Client Satisfaction Questionnaire (CSQ-8) instrument will be applied to evaluate satisfaction after implementation.

6.1.2. Feasibility Assessment

To evaluate the feasibility, the principal investigator will consider the following variables:

1. Recruitment of participants and sample characteristics.
2. Evaluation of data collection and results.
3. Evaluation of the acceptability of the intervention and study procedures and response rates.
4. Evaluation of resources and the ability to manage and implement the study and intervention.
5. Preliminary evaluation of participants responses to the intervention.
6. Level of progress of the participants in the sessions.

6.2 Secondary response measures: Validated measures for depression, anxiety, quality of life, distress tolerance, insomnia, emotion regulation, mindfulness skills, cognitive behavior theory skills, and suicide ideation will used at baseline, after the intervention, and four months after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students from the Universidad de los Andes, from different majors.
* Over 18 years.
* Able to read and speak Spanish.
* Availability of time to participate.

Exclusion Criteria:

* PHQ-9 score ≥ 15
* Active suicidality, defined as suicidal ideation, planning or attempts, or self-harming behavior in the last 12 months. The Columbia Suicidality Scale will be used to exclude students with a score ≥ 3.
* Who is undergoing psychiatric treatment for a serious condition, understood as psychotic pathology and/or substance abuse.
* History of hospital admission for psychiatric pathology in the last two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability Assessment | through study completion, an average of 1 year
  Acceptability will be evaluated by determining how this intervention program is received by students and the extent to which this intervention relates to the needs of this target population. The research team will develop an acceptability and satisfaction questionnaire and apply it to the intervention students.
Feasibility Assessment: Number of participants recruited | through study completion, an average of 1 year
  Initially, inclusion and exclusion criteria will be defined to ensure that participants are representatives of the target group. A tracking system will be implemented to monitor the number of people recruited.
Feasibility Assessment: Recruitment time for completion | through study completion, an average of 1 year
  A tracking system will be implemented to monitor the time needed to complete the recruitment process.
Feasibility Assessment: Evaluation of data collection and results. | through study completion, an average of 1 year
  Clear protocols will be established for data collection and analysis, ensuring accuracy and consistency. Statistical analyzes will be used to check the validity and reliability of the results.
Feasibility Assessment: Evaluation of the acceptability of the intervention | through study completion, an average of 1 year
  Surveys will be used to collect opinions and perceptions of participants about the intervention and the methods used.
Feasibility Assessment: Level of progress of the participants in the sessions. | through study completion, an average of 1 year
  The completion and the time needed for completion of each module of the intervention will be registered.
Client Satisfaction Questionnaire (CSQ-8) | through study completion, an average of 1 year
  It is an 8-item instrument validated in English and translated and validated into Spanish that measures general satisfaction with health services received in various populations. The answers are Likert-type with four options each. In addition, there is space to write down comments and suggestions. This instrument will be slightly adapted to questions oriented to the study context. The Customer Satisfaction Questionnaire has an internal consistency ranging between α=0.83 and α=0.93.
  Each item on the CSQ-8 is rated on a 4-point scale, generally ranging from 1 (low satisfaction) to 4 (high satisfaction). Therefore, the minimum possible score on the CSQ-8 is 8 (1 point on each of the 8 items), and the maximum score is 32 (4 points on each item).
  A higher score on the CSQ-8 indicates greater client satisfaction with the services received, which is considered a better outcome. In this context, a higher score is better, as it reflects a better customer perception of the service.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | through study completion, an average of 1 year
  It is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria from "0" (Never) to "3" (Almost Every Day). In Chile, it has been validated among people aged 20 years and over, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression Scale. In addition, it has construct validity and concurrent predictive validity with the The International Classification of Diseases, 10th Revision (CIE-10) criteria for depression. The interpretation is made by adding the total of the first nine questions: 0-4 points, without depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Generalized Anxiety Disorder (GAD-7) | through study completion, an average of 1 year
  GAD-7 was originally designed primarily as a screening and severity measure for generalized anxiety disorder, this instrument also has good performance characteristics for other common anxiety disorders: panic disorder, social anxiety disorder, and post-traumatic stress disorder. This consists of 7 questions. The score is calculated by assigning scores from 0 to 3 to response categories from "Never" to "Almost Every Day." It has been validated in Spanish, where a cut-off score of 10 showed adequate values of sensitivity (86.8%) and specificity (93.4%). The scale was significantly correlated with Hamilton Anxiety scal (HAM-A) (0.852, p < 0.001), Hospital Anxiety and Depression Scale (HADS ) (anxiety domain, 0.903, p < 0.001), and World Health Organization Disability Scale (WHO-DAS II) (0.696, p < 0.001). The GAD-7 total score for the seven items ranges from 0 to 21
PROMIS Global Health v1.2.: Patient-Reported Outcomes Measurement Information System (PROMIS) | through study completion, an average of 1 year
  It is an initiative of the National Institute of Health to develop measures that assess function and well-being in physical, mental, and social health domains. It has been translated into multiple languages and multiculturally validated. This instrument evaluates five areas: physical function, pain, fatigue, emotional stress, and social health. Four items are used to assess overall physical health, 3 of which use 5-category scales, and one item uses a 1-10 scale. Four items are used to determine global mental health, all using 5-category scales. Studies with the Spanish version of this instrument show good psychometric behavior.
Distress Tolerance Scale (DTS) | through study completion, an average of 1 year
  This instrument allows us to evaluate how people experience and endure distressing psychological states. The scale is constructed of 15 items, divided into four subscales that measure four factors: Tolerance (items 1, 3, and 5), understood as the perceived ability to handle strong emotions; Relief (items 2, 4, and 15), considered as "how relieved a person feels when they experience a strong emotion"; Evaluation (items 6, 7, 9, 10, 11 and 12), understood as the person's perceived ability to accept their strong emotions; and, Regulation (items 8, 13 and 14), understood as the effort that a person makes to manage their intense emotions openly. DTS is a scale designed to be self-administered that is answered using a type format.
Insomnia Severity Index (ISI) | through study completion, an average of 1 year
  It is a self-report instrument that measures the patient's perception of their insomnia. Its objective is subjective symptoms and consequences of insomnia. It was validated in English-speaking and Spanish-speaking populations. It is composed of 7 items, which gives a score that varies from 0 to 28, with clinical insomnia with 15 or more points.
The Emotion Regulation Questionnaire-Short Form (ERQ-S) | through study completion, an average of 1 year
  Is a 6-item self-report instrument of two common emotion regulation strategies: cognitive reappraisal (i.e., changing the way one thinks about a situation to change its emotional impact) and expressive suppression (i.e., inhibiting the expression behavior of emotion). It has a high level of reliability for each of the subscales: cognitive reappraisal subscale (α=0.87) and expressive suppression subscale (α=0.76).
  Each item on the ERQ-S is scored on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). In the short version of 6 items (3 for each subscale), the minimum possible score would be 6 (1 point in each of the 6 items) and the maximum would be 42 (7 points in each of the 6 items).
  In terms of interpretation of the scores, a higher score on each subscale indicates more frequent use of that specific emotion regulation strategy.
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | through study completion, an average of 1 year
  It is a 12-item scale that measures mindfulness in everyday situations. The items are scored from one to four on a Likert-type scale where 1 refers to "rarely or never" and 4 means "almost always." Therefore, the minimum possible score on the CAMS-R is 12, and the maximum score is 48. A higher score on the CAMS-R indicates a greater disposition or ability in mindfulness or full attention. It measures four subscales: attention, attentional focus on the present, awareness, and acceptance without judgment regarding thoughts and feelings in daily life. Despite measuring them in four factors, it analyzes them generally without separating them, offering a global score. According to different studies, internal consistency ranges from α=0.74 to α=0.80, with a negative correlation between depression and anxiety and a positive correlation with cognitive flexibility and well-being.
The Cognitive-behavioral Therapy Skills Questionnaire (CBTSQ) | through study completion, an average of 1 year
  Evaluates which components of Cognitive behavioral therapy (CBT) appear to be most active. This scale originally has 16 items that measures two skills: cognitive restructuring (CR) and behavioral activation (BA). Respondents rate each item on a 5-point Likert scale, from 1 (I don't do this) to 5 (I always do this). Both scales have good reliability (CR: α=0.88; BA: α=0.85). Two items refer to evaluating aspects related to a disease or treatment. Since cognitive-behavioral skills are evaluated in this study, these two items of the questionnaire are included, leaving an instrument of 14 items. In a study whose publication is under review with adolescents between 15 and 18 years old, using the 14-item instrument, it was found that the reliability was α=0.77 and ω=0.78 for BA and α=0, 80 and ω=0.81 for CR.
  The minimum score would be 14 and the maximum would be 70. A higher score on the CBTSQ indicates greater competence and use of cognitive behavioral therapy skills.
Columbia-Suicide Severity Rating Scale (C-SSRS) | through study completion, an average of 1 year
  The first 5 items explore the presence of suicidal ideation, intention, and planning and are assessed over the past month. The sixth item explores suicidal behavior either as preparation, initiation of a suicide attempt, or a suicide attempt itself in the last three months. Each item is answered Yes or No. It has been validated in an English-speaking population (range of internal reliability goes from α=0.73 to α=0.93) and a Spanish-speaking population (α=0.53). The total score range is from 0 to 6 points. According to the answers provided To the different items, the categories of severity of suicidal ideation are established: If the answer is "Yes" to item 1 and/or item 2 and "No" to all the other items, a slight risk is indicated. If the answer is "Yes" to item 2 and answer "Yes" only to item 3, it suggests that the risk is moderate. If the answer si "Yes" to item 2 and the answer is "Yes" to any of items 4, 5, and 6, it indicates that the risk is severe.
Mental Health History and Treatment: | through study completion, an average of 1 year
  Questions developed by the team will be used about history and previous mental health treatments and consultation with mental health services. Answers range from 0=No and 1=Yes.
Physical activity: | through study completion, an average of 1 year
  Three questions developed by the team will be used to meseaure physical activity (e.g., How many minutes the students practice any physical activity during the week or weekends).

IPD SHARING:
Plan to Share IPD: Yes
Data about primary and secondary outcomes without identifiable variables such as name, date of birth, or others.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study and until five years after the end of the study.
Access Criteria: Any researchers who ask the principal investigator fot secondary analysis, data anonymized.
URL: https://www.ismeuandes.cl/

REFERENCES:
- [Background] Hope V, Henderson M. Medical student depression, anxiety and distress outside North America: a systematic review. Med Educ. 2014 Oct;48(10):963-79. doi: 10.1111/medu.12512. PMID 25200017
- [Background] Valdes JM, Diaz FJ, Christiansen PM, Lorca GA, Solorza FJ, Alvear M, Ramirez S, Nunez D, Araya R, Gaete J. Mental Health and Related Factors Among Undergraduate Students During SARS-CoV-2 Pandemic: A Cross-Sectional Study. Front Psychiatry. 2022 May 31;13:833263. doi: 10.3389/fpsyt.2022.833263. eCollection 2022. PMID 35711588
- [Background] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Background] Preece DA, Petrova K, Mehta A, Gross JJ. The Emotion Regulation Questionnaire-Short Form (ERQ-S): A 6-item measure of cognitive reappraisal and expressive suppression. J Affect Disord. 2023 Nov 1;340:855-861. doi: 10.1016/j.jad.2023.08.076. Epub 2023 Aug 18. PMID 37597776
- [Background] Fernandez-Mendoza J, Rodriguez-Munoz A, Vela-Bueno A, Olavarrieta-Bernardino S, Calhoun SL, Bixler EO, Vgontzas AN. The Spanish version of the Insomnia Severity Index: a confirmatory factor analysis. Sleep Med. 2012 Feb;13(2):207-10. doi: 10.1016/j.sleep.2011.06.019. Epub 2011 Dec 14. PMID 22172961
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Hays RD, Schalet BD, Spritzer KL, Cella D. Two-item PROMIS(R) global physical and mental health scales. J Patient Rep Outcomes. 2017;1(1):2. doi: 10.1186/s41687-017-0003-8. Epub 2017 Sep 12. PMID 29757325
- [Background] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Background] Blatch-Jones AJ, Pek W, Kirkpatrick E, Ashton-Key M. Role of feasibility and pilot studies in randomised controlled trials: a cross-sectional study. BMJ Open. 2018 Sep 25;8(9):e022233. doi: 10.1136/bmjopen-2018-022233. PMID 30257847
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Segal ZV, Dimidjian S, Beck A, Boggs JM, Vanderkruik R, Metcalf CA, Gallop R, Felder JN, Levy J. Outcomes of Online Mindfulness-Based Cognitive Therapy for Patients With Residual Depressive Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):563-573. doi: 10.1001/jamapsychiatry.2019.4693. PMID 31995132
- [Background] Garland A, Weinfurt K, Sugarman J. Incentives and payments in pragmatic clinical trials: Scientific, ethical, and policy considerations. Clin Trials. 2021 Dec;18(6):699-705. doi: 10.1177/17407745211048178. PMID 34766524
- [Background] Murphy MJ, Newby JM, Butow P, Loughnan SA, Joubert AE, Kirsten L, Allison K, Shaw J, Shepherd HL, Smith J, Andrews G. Randomised controlled trial of internet-delivered cognitive behaviour therapy for clinical depression and/or anxiety in cancer survivors (iCanADAPT Early). Psychooncology. 2020 Jan;29(1):76-85. doi: 10.1002/pon.5267. Epub 2019 Nov 12. PMID 31659822
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Harrer M, Adam SH, Baumeister H, Cuijpers P, Karyotaki E, Auerbach RP, Kessler RC, Bruffaerts R, Berking M, Ebert DD. Internet interventions for mental health in university students: A systematic review and meta-analysis. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1759. doi: 10.1002/mpr.1759. Epub 2018 Dec 26. PMID 30585363
- [Background] Harrer M, Adam SH, Fleischmann RJ, Baumeister H, Auerbach R, Bruffaerts R, Cuijpers P, Kessler RC, Berking M, Lehr D, Ebert DD. Effectiveness of an Internet- and App-Based Intervention for College Students With Elevated Stress: Randomized Controlled Trial. J Med Internet Res. 2018 Apr 23;20(4):e136. doi: 10.2196/jmir.9293. PMID 29685870
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Bullis JR, Boe HJ, Asnaani A, Hofmann SG. The benefits of being mindful: trait mindfulness predicts less stress reactivity to suppression. J Behav Ther Exp Psychiatry. 2014 Mar;45(1):57-66. doi: 10.1016/j.jbtep.2013.07.006. Epub 2013 Jul 25. PMID 23994223
- [Background] Pacheco JP, Giacomin HT, Tam WW, Ribeiro TB, Arab C, Bezerra IM, Pinasco GC. Mental health problems among medical students in Brazil: a systematic review and meta-analysis. Braz J Psychiatry. 2017 Oct-Dec;39(4):369-378. doi: 10.1590/1516-4446-2017-2223. Epub 2017 Aug 31. PMID 28876408
- [Background] Lei XY, Xiao LM, Liu YN, Li YM. Prevalence of Depression among Chinese University Students: A Meta-Analysis. PLoS One. 2016 Apr 12;11(4):e0153454. doi: 10.1371/journal.pone.0153454. eCollection 2016. PMID 27070790
- [Background] Baader TM, Rojas CC, Molina JLF, Gotelli M V., Alamo CP, Fierro CF, et al. Diagnóstico de la prevalencia de trastornos de la salud mental en estudiantes universitarios y los factores de riesgo emocionales asociados. Rev Chil Neuropsiquiatr. 2014 Sep 1;52(3):167-76.
- [Background] Barrera-Herrera, A., & San Martín, Y. (2021). Prevalencia de Sintomatología de Salud Mental y Hábitos de Salud en una Muestra de Universitarios Chilenos. Psykhe, 30(1). https://doi.org/10.7764/psykhe.2019.21813
- [Background] Martínez, P., Jiménez-Molina, Á., Mac-Ginty, S., Martínez, V., & Rojas, G. (2021). Salud mental en estudiantes de educación superior en Chile: una revisión de alcance con meta-análisis. Terapia PsicolóGica (Impresa), 39(3), 405-426. https://doi.org/10.4067/s0718-48082021000300405).
- [Background] MacDonald HZ, Baxter EE. Mediators of the relationship between dispositional mindfulness and psychological well-being in female college students. Mindfulness. 2017;8:398-407.
- [Background] Mandal SP, Arya YK, Pandey R. Mindfulness, Emotion Regulation, and Subjective Well-Being: Exploring the Link. SIS Journal of Projective Psychology & Mental Health. 2017;24(1).
- [Background] Roemer L, Williston SK, Rollins LG. Mindfulness and emotion regulation. Current Opinion in Psychology. 2015;3:52-7.
- [Background] McDermott, R., & Dozois, D. J. A. (2019). A randomized controlled trial of Internet-delivered CBT and attention bias modification for early intervention of depression. Journal of Experimental Psychopathology, 10(2), 204380871984250. https://doi.org/10.1177/2043808719842502
- [Background] Santana VS, Gondim SMG. Regulação emocional, bem-estar psicológico e bem-estar subjetivo. Estudos de Psicologia (Natal). 2016;21:58-68.
- [Background] Giuliani NR, Berkman ET. Craving is an Affective State and Its Regulation Can Be Understood in Terms of the Extended Process Model of Emotion Regulation. Psychol Inq. 2015;26(1):48-53. doi: 10.1080/1047840X.2015.955072. No abstract available. PMID 25780321
- [Background] Küchler, A., Kählke, F., Vollbrecht, D., Peip, K., Ebert, D. D., & Baumeister, H. (2022). Effectiveness, Acceptability, and Mechanisms of Change of the Internet-Based Intervention StudiCare Mindfulness for College Students: a Randomized Controlled Trial. Mindfulness (New York. Print), 13(9), 2140-2154. https://doi.org/10.1007/s12671-022-01949-w
- [Background] Baader T, Molina JL, Venezian S, Rojas C, Farías R, Fierro-Freixenet C, et al. Validación y utilidad de la encuesta PHQ-9 (Patient Health Questionnaire) en el diagnóstico de depresión en pacientes usuarios de atención primaria en Chile. Revista chilena de neuro-psiquiatría. 2012;50(1):10-22.
- [Background] Simons JS, Gaher RM. The Distress Tolerance Scale: Development and Validation of a Self-Report Measure. Motivation and Emotion. 2005;29(2):83-102.
- [Background] Cardoso Ribeiro C, Gómez-Conesa A, Hidalgo Montesinos MD. Metodología para la adaptación de instrumentos de evaluación. Fisioterapia. 2010;32(6):264/70.
- [Background] Vázquez, F., Otero, P., López, L., Blanco, V., Torres, Á., & Dı́Az, O. (2018). La Prevención de la Depresión en Cuidadores a través de Multiconferencia Telefónica. Clínica Y Salud, 29(1), 14-20. https://doi.org/10.5093/clysa2018a2